CLINICAL TRIAL: NCT03271606
Title: The Clinical Study of ERAS Protocol in Video-assisted Mediastinal Surgery
Brief Title: ERAS in Video-assisted Mediastinal Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zs2017822
Record Dates: First submitted 2017-08-23; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERAS group (Experimental): The patients in this group receive enhanced measures perioperatively
  Interventions: Combination Product: ERAS
- Traditional group (Active Comparator): The patients in this group receive traditional measures perioperatively
  Interventions: Combination Product: Traditional measures

INTERVENTIONS:
Combination Product: ERAS — The investigators mainly used enhanced measures perioperatively in mediastinal surgery as these used in other surgery
  Arms: ERAS group
Combination Product: Traditional measures — The investigators mainly used traditional measures perioperatively in mediastinal surgery as these used in other surgery
  Arms: Traditional group

SUMMARY:
This is a single center, randomized,single blind study to investigate the effectiveness of enhanced recovery regimen (ERAS) in patients undergoing Video-assisted Mediastinal Surgery. And we also going to compare the effectiveness of ERAS with that of traditional regimen in these patients.

DETAILED DESCRIPTION:
Compare to traditional measures, the ERAS protocal mainly includes:Good preoperative visit, shorten the fast time, minimumal invasive surgery procedures, fewer opioids and early movements after surgery. These items have been successfully used in colon cancer surgery, and we thus plan to investigate the effectiveness of these measures in mediastinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients elective mediastinal surgery;
* BMI 18-30 kg/m2.

Exclusion Criteria:

* Patient refuse;
* ASA≥3;
* Patients allergic to used anesthetics (propofol,rocuronium), patients with liver and/or kidney and/or mental dysfunction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-02-23 (Estimated); Study Completion 2018-02-23 (Estimated)

PRIMARY OUTCOMES:
15-item quality of recovery scale (QoR-15) | At preoperative vist
  This scale mainly reflects the patient's status
15-item quality of recovery scale (QoR-15) | At 24 hours after surgery
  This scale mainly reflects the patient's status

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided